CLINICAL TRIAL: NCT04501783
Title: Randomized Open-label Multicenter Parallel-group Study of Efficacy and Safety of TL-FVP-t vs. Standard of Care Therapy in Patients With Mild to Moderate Coronavirus Disease (SARS-CoV-2/COVID-19)
Brief Title: Study of Efficacy and Safety of TL-FVP-t vs. SOC in Patients With Mild to Moderate COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TL-FVP-t-01
Record Dates: First submitted 2020-08-05; First posted 2020-08-06 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Severe acute respiratory syndrome coronavirus 2; 2019-nCoV; 2019 novel coronavirus; Respiratory disease; lung disease
MeSH Terms: conditions — COVID-19; Respiration Disorders; Lung Diseases | interventions — favipiravir; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TL-FVP-t (favipiravir) Treatment Arm (Experimental): Day 1: favipiravir 1800 mg BID plus Standard of Care (SOC); Days 2-10: 800 mg BID plus SOC.
  Interventions: Drug: Favipiravir; Drug: standard concomitant therapy
- Standard of Care Arm (Active Comparator): Standard of Care including etiotropic therapy according to MoH of Russian Federation Recomendations for COVID-19 (umifenovir + intranasal recombinant interferon alpha, or hydroxychloroquine, or chloroquine, or mefloquine in recomended regimen) up to10 days
  Interventions: Drug: Standard of care (SOC); Drug: standard concomitant therapy

INTERVENTIONS:
Drug: Favipiravir — TL-FVP-t will be administered orally
  Other Names: TL-FVP-t; Koronavir
  Arms: TL-FVP-t (favipiravir) Treatment Arm
Drug: Standard of care (SOC) — SOC will include standard etiotropic therapy (umifenovir + intranasal recombinant interferon alpha, or hydroxychloroquine, or chloroquine) according to MoH of Russian Federation recomendations for COVID-19
  Arms: Standard of Care Arm
Drug: standard concomitant therapy — Standard of care according to MoH of Russian Federation recomendation for COVID-19

SUMMARY:
Randomized open-label multicenter parallel-group study of efficacy and safety of TL-FVP-t vs. standard of care therapy in patients with mild to moderate coronavirus disease (SARS-CoV-2/COVID-19)

DETAILED DESCRIPTION:
This was an open label, randomized, controlled, multicenter Phase 3 study of TL-FVP-t in outpatients and inpatients with mild to moderate COVID-19. After stratification by the severity of their disease (mild or moderate), age (18-44 or ≥ 45 years) and CT severity subjects were randomized at a rate of 2:1 to receive either TL-FVP-t + standard concomitant therapy or standard ethiptropic therapy (standard of care - SOC) including standard concomitant therapy. Standard ethiptropic therapy according to MoH of Russian Federation included umifenovir + intranasal recombinant interferon alpha, hydroxichloroquine, or chloroquine.

The dose regimen was the following: TL-FVP-t at a dose of 1800 mg BID on the Day 1 followed by 800 mg BID during the next 9 days. The study included the period of therapy (10 days) and follow-up period (18 days).

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form signed.
2. Males and females aged 18-60 years;
3. Diagnosis of coronavirus disease caused by SARS-CoV-2 (COVID-19) in a mild or moderate form (without respiratory failure).
4. Duration of infection symptoms shall be no more than 6 days before randomization.
5. SARS-CoV-2 infection should be verified by PCR at the screening.
6. Ability to follow the protocol and fulfill all the clinical study procedures.
7. Ability and willingness of the subjects and their sexual partners with retained childbearing potential to use reliable contraception methods throughout the study and for 3 months after the treatment completion.
8. Willingness not to take alcohol throughout the study.

Exclusion Criteria:

1. Age < 18 and > 60 years.
2. Any etiotropic therapy of coronavirus SARS-CoV-2 (COVID-19) infection prior to the study.
3. Moderate infection with respiratory failure, severe or extremely severe SARS-CoV-2 (COVID-19) disease.
4. Respiratory failure (RR > 30/min, SpO2 ≤ 93 %) or the need for mechanical ventilation at the screening.
5. Decreased level of consciousness (disorientation of place, time and personality), agitation at the screening.
6. Unstable hemodynamics (systolic BP < 100 mm Hg or diastolic BP < 60 mm Hg) found at the screening.
7. Subtotal diffuse ground-glass induration of pulmonary tissue and pulmonary consolidation combined with reticular changes; involvement of ≥ 75 % of lung parenchyma; hydrothorax (CT findings corresponding to ≥ CT-4 according to Department of Health of Moscow guidelines).
8. Presence of comorbidities:

   1. moderate or severe chronic obstructive pulmonary disease or asthma;
   2. severe chronic cardiovascular disorders (arrhythmia or conduction disorders, implanted pacemaker device, myocardial infarction or unstable angina in the medical history, heart failure);
   3. immunocompromised subjects (HIV, cancer, autoimmune diseases, immunodepressant therapy);
   4. severe obesity (body mass index [BMI] ≥ 40);
   5. diabetes mellitus;
   6. chronic renal failure;
   7. chronic moderate or severe hepatic disorders.
9. Any of the following abnormal laboratory tests at the screening: AST or ALT level > 2.5 x upper normal level (UNL), platelet count < 50х109/L.
10. Any history findings which, in the investigator's opinion, may complicate the interpretation of the study results or generate an additional risk for the subject due to his/her participation in the study.
11. More than 2 CT diagnostic procedures within the last 6 months prior to randomization (except for chest CT no earlier than 4 days prior to enrollment).
12. The subject takes the products significantly inhibiting CYP28С, and administration those products cannot be interrupted for the study duration.
13. Malabsorption syndrome or another clinically relevant gastrointestinal disease which may affect the study product absorption (uncontrollable vomiting, diarrhea, ulcerative colitis, etc.).
14. Pregnancy or breast-feeding; women with probable pregnancy at the screening, those planning to conceive during the study.
15. Known (from the history) or suspected alcohol or psychotropic drug abuse; medicinal or illicit drug addiction.
16. Mental disorders including those in the medical history.
17. Condition or disease which, according to the investigator or medical monitor, will compromise the subject's safety or affect assessment of the study product safety.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
Time to clinical improvement | through Day 28
  To determine the effect of TL-FVP-t vs. SOC on time to clinical improvement. The clinical improvement is defined as reduction on at least 1 score of patient clinical status according to WHO 8-category Ordinal Scale for Clinical Improvement compared to screening
Time to viral clearance | through Day 28
  To determine the effect of TL-FVP-t vs. SOC on time to viral clearance of SARS-CoV-2 virus as measured by PCR in oropharyngeal sampling

SECONDARY OUTCOMES:
Rate of clinical improvement at separate time points | Day 7
  To determine the effect of TL-FVP-t vs. SOC on proportion of subjects (%) with clinical improvement according to WHO 8-category Ordinal Scale for Clinical Improvement
Rate of viral clearance at separate time points | Days 5 and 7
  To determine the effect of TL-FVP-t vs. SOC on a proportion of subjects (%) with viral clearance of SARS-CoV-2 virus as measured by PCR in oropharyngeal sampling at separate time points
Time to body temperature normalization | through Day 28
  To determine the effect of TL-FVP-t vs. SOC on time to body temperature normalization determined as body temperature < 37°C without antipyretics for at least 48 hours.
Rate of resolution of lung changes on CT | Day 14
  To determine the effect of TL-FVP-t vs. SOC on a proportion of subjects (%) with resolution of lung changes on CT
Rate of adverse drug reactions (ADR) and serious ADR | through Day 28
  To determine the effect of TL-FVP-t vs. SOC on a proportion of subjects (%) with ADR and serious ADR
Rate of severe ADR | through Day 28
  To determine the effect of TL-FVP-t vs. SOC on a proportion of subjects (%) with severe ADR
Rate therapy termination due to ADR | through Day 28
  To determine the effect of TL-FVP-t vs. SOC on a proportion of subjects (%) discontinued therapy due ADR

CONTACTS AND LOCATIONS:
Locations (10):
- Russia (10):
  - Medical center LLC "Neuroprofi", Korolyov
  - Federal budgetary institution of science "Central Research Institute of Epidemiology" of Russian Federal Supervision Service for Consumer Rights Protection and People's Welfare, Moscow
  - Medical centers JSC "Medsi Group of Companies", Moscow
  - State budgetary institution of health care of the city of Moscow "City Clinical Hospital №52 of the Moscow City Healthcare Department", Moscow
  - State budgetary institution of health care of the city of Moscow "City Clinical Hospital №67 n.a. LA Vorokhobova of the Moscow City Healthcare Department", Moscow
  - State budgetary institution of health care of the city of Moscow "Infectious Diseases Clinical Hospital №1 of the Moscow City Healthcare Department", Moscow
  - Medical center LLC "Medical Center Eco-safety", Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "City Hospital No. 40 of the Kurortny District", Saint Petersburg
  - Budgetary healthcare institution of the Voronezh region "Voronezh Regional Clinical Hospital No. 1", Voronezh
  - State Budgetary Healthcare Institution of the Moscow Region "Zhukovskaya City Clinical Hospital"., Zhukovskiy

IPD SHARING:
Plan to Share IPD: No